CLINICAL TRIAL: NCT03545893
Title: A Pilot Randomized Trial of Opioids Versus Nonopioids for Pain Control After Osmotic Dilator Placement for Abortion Care
Brief Title: Overnight Pain Treatment Investigating Opioids vs. Nonopioids
Acronym: OPTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 829723
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Abortion Second Trimester
MeSH Terms: interventions — Ibuprofen; Oxycodone; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen 600 mg
- Ibuprofen + Oxycodone (Active Comparator)
  Interventions: Drug: Ibuprofen 600 mg; Drug: OxyCODONE 5 Mg Oral Tablet

INTERVENTIONS:
Drug: Ibuprofen 600 mg — Ibuprofen 600mg prescription, to be taken 1 tablet as needed every 6 hours for pain.
Drug: OxyCODONE 5 Mg Oral Tablet — Oxycodone 5mg Oral Tablet prescription, to be taken 1-2 tablets as needed every 6 hours for pain.
  Arms: Ibuprofen + Oxycodone

SUMMARY:
The purpose of this study is to compare maximum pain scores between patients seeking induced abortion and requiring cervical preparation with osmotic dilators. Patients will be randomized to receive prescription for ibuprofen alone or to receive prescription for ibuprofen + oxycodone for overnight pain management after cervical preparation with osmotic dilators. Data collected in-person and through a text-messaging platform.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking women
* 18 years or older
* Access to cell phone with text-messaging capability/data
* Receiving cervical preparation for induced abortion
* Able to complete baseline survey on smartphone/tablet at screening visit

Exclusion Criteria:

* History of opioid or alcohol abuse
* Contraindications or allergy to ibuprofen
* Contraindications or allergy opioid medications
* Seeking uterine evacuation for premature preterm rupture of membranes or advanced - cervical dilation or intrauterine fetal demise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibuprofen | Ibuprofen + Oxycodone
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Ibuprofen + Oxycodone | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (7.7) | 30.9 (8.6) | 30.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 18 | 37
  White | 11 | 10 | 21
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Maximum Pain Score
Description: Numerical Rating Scale (NRS) pain score (scale range 0-10, with a 0 meaning "no pain" and 10 meaning the "worst possible pain")
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen | Ibuprofen + Oxycodone
Number analyzed (Participants) | 35 | 35
score on a scale | 4.66 (2.86) | 6.51 (2.50)

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Ibuprofen | Ibuprofen + Oxycodone
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 35/35 | 35/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=35) | Ibuprofen + Oxycodone (N=35)
Nausea (Gastrointestinal disorders) | 11 (11) | 18 (18)
Uterine Cramping (Reproductive system and breast disorders) | 29 (29) | 29 (29)
Vaginal spotting (Reproductive system and breast disorders) | 18 (18) | 22 (22)
Vaginal bleeding (Reproductive system and breast disorders) | 6 (6) | 12 (12)
Uterine pain (Reproductive system and breast disorders) | 4 (4) | 6 (6)
Dizziness (Nervous system disorders) | 2 (2) | 6 (6)
Drowsiness (Nervous system disorders) | 2 (2) | 7 (7)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT03545893/Prot_SAP_000.pdf